CLINICAL TRIAL: NCT04668742
Title: A Clinical, Controlled, Randomized Trial to Evaluate the Efficacy and Safety of the New Dynatraq Invention Device to Prevent Complications Associated With Tracheostomy Tubes in Mechanically Ventilated Patients: " Dynatraq-2 Study "
Brief Title: Efficacy and Safety of the DYNAtraq Device to Prevent Complications in Tracheostomy in Mechanically Ventilated Patients
Acronym: DYNAtraq
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Cardiovascular de Colombia (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government); Plasticos de Santander Ltda PLADESAN (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 656677758319
Record Dates: First submitted 2020-11-23; First posted 2020-12-16 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Tracheostomy; Mechanical Ventilation Complication
Keywords: tracheostomy; airway; complications

STUDY DESIGN:
Who Masked: Investigator
Masking Description: masking of the intervention and control groups in the statistical analysis of the data, which will be represented as group 0 and 1, without identifying whether they are control or intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: DYNAtraq - tracheostomy fixation device (Experimental): Use of DYNatraq installed in chest with skin adhesive and fixed to tracheostomy tube
  Interventions: Device: DYNAtraq
- Arm 2: Usual management of tracheostomy (No Intervention): No interventions will be used additional to usual management

INTERVENTIONS:
Device: DYNAtraq — Tracheostomy alignment with DYNAtraq
  Other Names: tracheostomy fixation device
  Arms: Arm 1: DYNAtraq - tracheostomy fixation device

SUMMARY:
Although tracheostomy is a common technique in Intensive Care Units (ICU), its complications can be frequent (between 5% to 40%). Inadequate fixation could favor decannulation, as well as incorrect alignment of the tracheostomy with respect to the tracheal axis could favor the appearance of tissue alterations such as ulcers, bleeding or fistulas, as well as obstruction of the ventilatory obstruction. Having a device that is effective in fixation and alignment could help in reducing tracheostomy complications, so this study aims to evaluate the effect and safety of a fixation device for tracheostomy through a randomized clinical trial.

DETAILED DESCRIPTION:
Introduction: Tracheostomy is one of the most frequently required surgical techniques for the management of hospitalized patients in Intensive Care Units (ICU). This procedure is justified to facilitate the improvement of the patient, facilitate early rehabilitation, reduce sedation and analgesia requirements, and reduce the length of stay in the ICU and the days of mechanical ventilation (MV). However, tracheostomy is associated with various complications, from mispositioning and accidental decannulation, to hemoptysis, tracheal fistulas, air leaks, and ventilatory difficulties. In a pre-post quasi-experimental study where the effect of the DYNAtraq technological innovation device on tracheostomy fixation and alignment was evaluated, it was found that it can correct 83% of cases, which contrasts with only 2% when they did not have the device. (p <0.01). This previous study allowed us to conclude that technological innovation through DYNAtraq is pertinent, relevant and effective to correct the position of tracheostomy tubes in patients hospitalized in the ICU and under mechanical ventilation.

Objective: To evaluate the efficacy and safety of the DYNAtraq medical device to keep tracheostomy tubes in correct alignment and fixation in adult patients with tracheostomy hospitalized in the ICU and under invasive mechanical ventilation.

Methodology: Randomized, controlled clinical trial (two-parallel arm), assigned in a 1: 1 ratio, in a sample of 74 patients mechanically ventilated in intensive care unit (37 in intervention group and 37 patients in control group). This study is conducted in two centers for intensive care patients in two Colombian cities and

The patients randomized to the intervention group will have the external fixation system for the tracheostomy installed, which is a non-invasive plastic device, from the start of the tracheostomy to ventilatory weaning. Patients in the control group will receive the usual management of the tracheostomy given in ICU. To evaluate alignment , the cephalo-caudal (C-C) and lateral-lateral (L-L) angles will be evaluated through photographs and analyzed with the SAPO application. The mean values of the angles were obtained in degrees and their 95% confidence intervals. Angular means were compared using the paired Student's t test.

Expected Results: The DYNAtraq device is expected to be effective in improving the proper fixation, orientation, and alignment of the tracheostomy tube in mechanically ventilated patients, reducing the complications of lacerations, bleeding, decannulation, and respiratory infectious complications.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Indication for a tracheostomy
* Signature of informed consent

Exclusion criteria:

* Mediastinitis
* Open chest
* Chest skin infection /burns anterior region of the thorax
* Patients requiring reanimation
* Active phase of COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Presence of mis-alignment of tracheostomy tube | 72 hours after tracheostomy installation
  Deviation from 95° angle of tracheostomy tube (cephalo-caudal (C-C) and lateral-lateral (L-L) angles) No evidence of alignment of tube though bronchoscopy

SECONDARY OUTCOMES:
Presence of complications of tracheostomy | 72 hours after tracheostomy installation
  Evidence of any complication due to tracheostomy (infections, bleeding, extubation, death)

OTHER OUTCOMES:
Presence of skin lesion | 72 hours after tracheostomy installation
  Safety of the device in skin (adhesive)

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Orozco-Levi, Ph.D, Principal Investigator — Fundacion Cardiovascular de Colombia- Hospital internacional de Colombia
Locations (1):
- Hospital Internacional de Colombia, Piedecuesta, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: No